CLINICAL TRIAL: NCT05511935
Title: Testing Preliminary Effectiveness of a Training to Support CHWs Outreach on Dental to African American Caregivers
Acronym: GRIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KDH Research & Communication (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-02-04; 1R43MD016352 (NIH)
Record Dates: First submitted 2022-08-16; First posted 2022-08-23 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Oral Health; Child; Adolescents; Self Efficacy; Intention; Health Literacy; African Americans; Poverty; Community Health Workers; Attitude; Knowledge
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exposed to GRIN training (Experimental): participates in the intervention
  Interventions: Other: professional development training for CHWs on dental health (GRIN)
- control/unexposed (No Intervention): no intervention

INTERVENTIONS:
Other: professional development training for CHWs on dental health (GRIN) — multi module online training
  Arms: exposed to GRIN training

SUMMARY:
Two arm study, experimental and control, to explore the impact of an online training program to help community health workers conduct effective outreach to support the dental health of African American youth via their caregivers.

DETAILED DESCRIPTION:
The investigators will use a randomized, two-group, pretest/posttest design to test the efficacy of the GRIN prototype and explore the following research question: To what extent does exposure to the GRIN prototype relate to positive changes in CHWs' knowledge, attitudes and beliefs, perceived self-efficacy, and intent to conduct oral health care outreach to low-income Black guardians? The community-driven nature of the project will ground the evaluation in the principles of an equitable evaluation that incorporates a racial equity lens. An equitable evaluation is "an approach that addresses the dynamics and practices that have historically undervalued the voices, knowledge, expertise, capacity, and experiences of all evaluation participants and stakeholders, particularly people of color and other marginalized groups." This approach "requires that evaluators engage in a process of ongoing self-reflection and adjustment, including a willingness to question and adapt traditional evaluation methods in response to stakeholder input." Working with communities to reflect the specific needs of their constituents, investigators will develop and enhance collaborations that leverage stakeholder expertise; minimize counter-productive duplications of services and resource expenditure; and create empowered opportunities for CHWs to conduct outreach with low-income Black guardians. The PI, with input from the SC, will develop necessary research materials, including the recruitment protocols, evaluation instrumentation, and human subjects consent materials, which then be reviewed against an equitable evaluation checklist, obtaining input on revisions from community members where needed. The PI will also outline the appropriate statistical analysis methods. All procedure documents will be reviewed by the KDHRC Institutional Review Board before the evaluation launch.

The investigators will recruit participants through evaluation partners who will disseminate the study information to CHWs via electronic notifications and flyers. Evaluation partners include National Association of Community Health Workers (NACHW) and the University of Southern Mississippi College of Nursing and Health Professionals (see Letters of Support for more details). The notification will provide information about the goal of the study, participant eligibility, and a link to an interest and eligibility form. Once a potential participant completes the interest and eligibility form and s/he is eligible for the project, they will receive a link to a consent form located on a secure online platform.

CHWs will be randomly assigned to the intervention or control group after consent and enrollment in the study. All participants will complete an online pretest survey. The intervention group will be exposed to GRIN and will complete an online posttest survey two weeks after completing the GRIN modules. The control group participants will not be exposed to the GRIN program and will complete a posttest two weeks after completing the pretest. Participant responses to pretest and posttest survey measures will be linked using non-personal identifiers.

The investigators will download and export the data from SurveyGizmo into an encrypted Excel file and import the raw data into STATA. The investigators will match the pretest and posttest responses using the random assigned identifiers and conduct analyses to test for the effect of GRIN exposure on changes in CHWs' knowledge, attitudes and beliefs, self-efficacy, and intentions to conduct pediatric oral health care outreach to low-income Black guardians. The a priori feasibility criterion is: Statistically significant differences between pretest and posttest knowledge and self-efficacy measures among the intervention group participants.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old.
* Must self-identify as a community health worker.
* Must conduct outreach to Black parents of children and adolescents.
* Must have six months of field experience. KDHRC defines "field experience" as conducting outreach activities in their community, for example, working with clients in a clinic, conducting home visits, or educating clients at health fairs or community events
* Must be an active CHW. KDHRC defines "active" as conducting outreach activities, such as working with clients in a clinic, conducting home visits, or educating clients at health fairs or community events, in the last six months.
* Must have Internet access either at home or at work to access the the GRIN virtual education session and/or online surveys.

Exclusion criteria:

-None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Twombly, PhD, Study Chair — KDH Research & Communication
Locations (1):
- KDH Research & Communication, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited participants from AHECS in MD, PA, TX, and the National Association of Community Health Workers.
Period: Overall Study
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Started | 71 | 72
Completed | 62 | 45
Not Completed | 9 | 27
Not completed — Lost to Follow-up | 9 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exposed to GRIN Training | Control/Unexposed | Total
Number analyzed (Participants) | 62 | 45 | 107
Age, Categorical [Count of Participants; unit: Participants] — Population: Two control participants left this answer blank.
  Participants
    number analyzed (Participants) | 62 | 43 | 105
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 61 | 43 | 104
    >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One treatment and two control participants left this question blank.
  Participants
    number analyzed (Participants) | 61 | 43 | 104
    Female | 57 | 35 | 92
    Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two treatment and three control group participants left this question blank.
  Participants
    number analyzed (Participants) | 60 | 42 | 102
    Hispanic or Latino | 11 | 16 | 27
    Not Hispanic or Latino | 48 | 26 | 74
    Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 23 treatment and 2 control left this question blank.
  Participants
    number analyzed (Participants) | 39 | 43 | 82
    American Indian or Alaska Native | 0 | 2 | 2
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 19 | 16 | 35
    White | 15 | 14 | 29
    More than one race | 1 | 7 | 8
    Unknown or Not Reported | 3 | 3 | 6
Highest education level completed [Count of Participants; unit: Participants] — Population: 2 control participants left this question blank
  Participants
    number analyzed (Participants) | 62 | 43 | 105
    Highschool diploma/GED | 1 | 5 | 6
    Some college | 20 | 9 | 29
    College degree | 33 | 22 | 55
    Master's degree | 5 | 5 | 10
    Professional degree | 3 | 2 | 5
Length of time serving as a community health worker [Count of Participants; unit: Participants] — Population: Two participants from each group left this question blank.
  Participants
    number analyzed (Participants) | 60 | 43 | 103
    Less than 6 months | 6 | 5 | 11
    6 to 11 months | 7 | 7 | 14
    1 to 2 years | 18 | 13 | 31
    3 to 4 years | 9 | 12 | 21
    5 or more years | 20 | 6 | 26
Paid or volunteer CHW position [Count of Participants; unit: Participants] — Population: One treatment and two control participants left this question blank.
  Participants
    number analyzed (Participants) | 61 | 43 | 104
    Paid | 55 | 33 | 88
    Volunteer | 2 | 3 | 5
    Both paid and volunteer | 4 | 7 | 11
Number of hours of community health worker training [Count of Participants; unit: Participants] — Population: One treatment and three control participants left this question blank.
  Participants
    number analyzed (Participants) | 61 | 42 | 103
    None | 2 | 0 | 2
    1 to 5 hours | 3 | 0 | 3
    6 to 10 hours | 2 | 1 | 3
    11 to 15 hours | 4 | 1 | 5
    16+ hours | 50 | 40 | 90
Previously received training about oral health for children/adolescents [Count of Participants; unit: Participants] — Population: One treatment and two control participants left this question blank.
  Participants
    number analyzed (Participants) | 61 | 43 | 104
    Yes | 15 | 13 | 28
    No | 43 | 28 | 71
    Don't know | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Pretest Score
Description: We asked participants 12 multiple choice knowledge questions related to oral health which we averaged to create a composite knowledge score for each participant ranging from 0 to 100. A score of 0 meant a participant got zero questions correct while a score of 100 meant a participant got all questions correct. We averaged these composite scores across all participants for both groups to create mean scores ranging from 0 to 100, the higher the score the more questions participants answered correctly.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Number analyzed (Participants) | 62 | 45
score on a scale | 64.92 (20.03) | 66.67 (17.04)
Statistical Analysis 1: Comparison: Exposed to GRIN Training vs Control/Unexposed; Test type: Superiority; p = 0.64, t-test, 2 sided; Mean Difference (Final Values) = 1.75, 95% CI 2-sided [-5.57 to 9.06], Standard Error of Mean 3.69

2. Primary Outcome: Attitudes Pretest Score
Description: We asked all participants seven Likert-type scale questions about attitudes towards conducting oral health outreach. Each answer choice rating ranged from 1 to 10, with higher ratings representing higher perceptions of oral health outreach importance. We averaged ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest score and 10 being the highest. Higher score means better outcome. Then, we averaged these composite scores for each group.
Time Frame: Baseline
Population: 11 treatment and 3 control participants did not answer all of the individual outcome questions and thus did not have composite scores included in the final average scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Number analyzed (Participants) | 51 | 42
score on a scale | 8.46 (0.88) | 8.60 (0.85)
Statistical Analysis 1: Comparison: Exposed to GRIN Training vs Control/Unexposed; Test type: Superiority; p = 0.47, t-test, 2 sided; Mean Difference (Final Values) = 1.30, 95% CI 2-sided [-2.28 to 4.89], Standard Error of Mean 1.81

3. Primary Outcome: Self-efficacy Pretest Score
Description: We asked all participants 10 Likert-type scale questions related to perceived self-efficacy with conducting oral health outreach. Each rating ranged from 1 to 10, with higher ratings representing higher perceptions of confidence in providing oral health outreach. We averaged ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, averaged these composite scores for both groups.
Time Frame: Baseline
Population: 11 treatment and 2 control participants did not answer all of the individual outcome questions and thus did not have composite scores included in the final average scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Number analyzed (Participants) | 51 | 43
score on a scale | 8.16 (1.90) | 7.93 (2.22)
Statistical Analysis 1: Comparison: Exposed to GRIN Training vs Control/Unexposed; Test type: Superiority; p = 0.59, t-test, 2 sided; Mean Difference (Final Values) = -2.33, 95% CI 2-sided [-10.77 to 6.11], Standard Error of Mean 4.25

4. Primary Outcome: Intentions Pretest Score
Description: We asked all participants five Likert-type scale questions related to their intentions to conduct oral health outreach. Each rating ranged from 1 to 10, with higher ratings representing higher perceived likelihood of providing oral health outreach in the future. We averaged ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, averaged these composite scores for each group.
Time Frame: Baseline
Population: 10 treatment and 8 control participants did not answer all of the individual outcome questions and thus did not have composite scores included in the final average scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Number analyzed (Participants) | 52 | 37
score on a scale | 7.39 (2.32) | 7.23 (2.89)
Statistical Analysis 1: Comparison: Exposed to GRIN Training vs Control/Unexposed; Test type: Superiority; p = 0.77, t-test, 2 sided; Mean Difference (Final Values) = -1.61, 95% CI 2-sided [-12.61 to 9.38], Standard Error of Mean 5.53

5. Primary Outcome: Knowledge Posttest Score
Description: We asked participants 12 multiple choice knowledge questions related to oral health which we averaged to create a composite knowledge score for each participant ranging from 0 to 100. A score of 0 meant a participant got zero questions correct while a score of 100 meant a participant got all questions correct. We averaged these composite scores across all participants for both groups to create mean scores ranging from 0 to 100. Higher scores mean better outcome.
Time Frame: Posttest (2 weeks after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Number analyzed (Participants) | 62 | 45
score on a scale | 79.44 (13.97) | 67.22 (15.83)
Statistical Analysis 1: Comparison: Exposed to GRIN Training vs Control/Unexposed; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -12.21, 95% CI 2-sided [-17.95 to -6.47], Standard Error of Mean 2.89

6. Primary Outcome: Attitudes Posttest Score
Description: We asked all participants seven Likert-type scale questions about attitudes towards conducting oral health outreach. Each rating ranged from 1 to 10, with higher ratings representing higher perceptions of oral health outreach importance. We averaged ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, averaged these composite scores for each group.
Time Frame: Posttest (2 weeks after baseline)
Population: 16 treatment and 6 control participants did not answer all of the individual outcome questions and thus did not have composite scores included in the final average scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Number analyzed (Participants) | 46 | 39
score on a scale | 8.45 (0.99) | 8.62 (0.67)
Statistical Analysis 1: Comparison: Exposed to GRIN Training vs Control/Unexposed; Test type: Superiority; p = 0.39, t-test, 2 sided; Mean Difference (Final Values) = 1.62, 95% CI 2-sided [-2.10 to 5.34], Standard Error of Mean 1.87

7. Primary Outcome: Self-efficacy Posttest Score
Description: We asked all participants 10 Likert-type scale questions related to perceived self-efficacy with conducting oral health outreach. Each rating ranged from 1 to 10, with higher ratings representing higher perceptions of confidence in providing oral health outreach. We averaged ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, averaged these composite scores for each group.
Time Frame: Posttest (2 weeks after baseline)
Population: 3 treatment and 5 control participants did not answer all of the individual outcome questions and thus did not have composite scores included in the final average scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Number analyzed (Participants) | 59 | 40
score on a scale | 9.36 (1.08) | 8.48 (1.75)
Statistical Analysis 1: Comparison: Exposed to GRIN Training vs Control/Unexposed; Test type: Superiority; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = -8.88, 95% CI 2-sided [-14.52 to -3.24], Standard Error of Mean 2.84

8. Primary Outcome: Intentions Posttest Score
Description: as for outcome 4
Time Frame: Posttest (2 weeks after baseline)
Population: 6 treatment and 5 control participants did not answer all of the individual outcome questions and thus did not have composite scores included in the final average scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Number analyzed (Participants) | 56 | 40
score on a scale | 8.38 (1.77) | 8.10 (2.20)
Statistical Analysis 1: Comparison: Exposed to GRIN Training vs Control/Unexposed; Test type: Superiority; p = 0.49, t-test, 2 sided; Mean Difference (Final Values) = -2.84, 95% CI 2-sided [-10.90 to 5.23], Standard Error of Mean 4.06

9. Secondary Outcome: Satisfaction at Posttest Score
Description: We asked only the intervention group participants five Likert-type scale questions related to their satisfaction with the GRIN intervention. Each rating ranged from 1 to 5, with higher scores representing higher satisfaction with the GRIN intervention. We averaged ratings from each question to create an average composite rating for each intervention participant, then averaged these scores across the intervention group. Scores ranged from 1 to 5, with higher scores meaning better satisfaction/outcome.
Time Frame: Baseline (2 weeks after baseline)
Population: 28 treatment participants did not answer all of the individual satisfaction outcome questions and thus did not have composite scores included in the final average score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training
Number analyzed (Participants) | 34
score on a scale | 4.49 (0.46)

10. Post Hoc Outcome: Change in Knowledge Scores From Pretest to Posttest
Description: At both pretest and posttest, we asked all participants the same 12 multiple choice knowledge questions related to oral health, which we averaged to create a composite knowledge score for each participant ranging from 0 to 100. A score of 0 meant a participant got zero questions correct while a score of 100 meant a participant got all questions correct. We averaged these composite scores across all participants for both groups to create mean scores. We then subtracted pretest scores from posttest scores and averaged these changes for all participants as the dependent variable in multiple regression. Higher scores mean higher gains from baseline to posttest. We used group assignment (intervention or treatment) as the main independent variable while controlling for participant baseline characteristics and demographics.
Time Frame: From baseline to posttest (2 weeks)
Population: Lower numbers were analyzed for both groups in the regression analyses due to missing data in the control variables.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Number analyzed (Participants) | 31 | 36
score on a scale | 14.52 (17.98) | 0.56 (13.22)
Statistical Analysis 1: Comparison: Exposed to GRIN Training vs Control/Unexposed; Test type: Superiority; p = 0.15, Regression, Linear; Slope = 7.71, 95% CI 2-sided [-2.92 to 18.35], Standard Error of Mean 5.28

11. Post Hoc Outcome: Change in Attitude Scores From Pretest to Posttest
Description: We asked all participants seven Likert-type scale questions about attitudes towards conducting oral health outreach. Each rating ranged from 1 to 10, with higher ratings representing higher perceptions of oral health outreach importance. We averaged ratings from each question to create an average composite rating for each participant, then averaged these composite scores for both groups. We then subtracted pretest scores from posttest scores and averaged these changes for all participants as the dependent variable in multiple regression. Higher scores mean higher gains from baseline to posttest. We used group assignment (intervention or treatment) as the main independent variable while controlling for participant baseline characteristics and demographics.
Time Frame: From baseline to posttest (2 weeks)
Population: Lower numbers were analyzed for both groups in the regression analyses due to missing data in the control variables.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Number analyzed (Participants) | 23 | 29
score on a scale | -0.07 (1.27) | 0.05 (0.86)
Statistical Analysis 1: Comparison: Exposed to GRIN Training vs Control/Unexposed; Test type: Superiority; p = 0.92, Regression, Linear; Slope = 0.43, 95% CI 2-sided [-8.13 to 8.99], Standard Error of Mean 4.19

12. Post Hoc Outcome: Change in Self-efficacy Scores From Pretest to Posttest
Description: We asked all participants 10 Likert-type scale questions related to perceived self-efficacy with conducting oral health outreach. Each rating ranged from 1 to 10, with higher ratings representing higher perceptions of confidence in providing oral health outreach. We averaged ratings from each question to create an average composite rating for each participant, then averaged these composite scores for both groups. We then subtracted pretest scores from posttest scores and averaged these changes for all participants as the dependent variable in multiple regression. Higher scores mean higher gains from baseline to posttest. We used group assignment (intervention or treatment) as the main independent variable while controlling for participant baseline characteristics and demographics.
Time Frame: From baseline to posttest (2 weeks)
Population: Lower numbers were analyzed for both groups in the regression analyses due to missing data in the control variables.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Number analyzed (Participants) | 26 | 29
score on a scale | 1.14 (0.24) | 0.46 (1.00)
Statistical Analysis 1: Comparison: Exposed to GRIN Training vs Control/Unexposed; Test type: Superiority; p = 0.20, Regression, Linear; Slope = 7.66, 95% CI 2-sided [-4.17 to 19.49], Standard Error of Mean 5.81

13. Post Hoc Outcome: Change in Intentions Scores From Pretest to Posttest
Description: We asked all participants five Likert-type scale questions related to their intentions to conduct oral health outreach. Each rating ranged from 1 to 10, with higher ratings representing higher perceived likelihood of providing oral health outreach in the future. We averaged ratings from each question to create an average composite rating for each participant, then averaged these composite scores for both groups. We then subtracted pretest scores from posttest scores and averaged these changes for all participants as the dependent variable in multiple regression. Higher scores mean higher gains from baseline to posttest. We used group assignment (intervention or treatment) as the main independent variable while controlling for participant baseline characteristics and demographics.
Time Frame: From baseline to posttest (2 weeks)
Population: Lower numbers were analyzed for both groups in the regression analyses due to missing data in the control variables.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposed to GRIN Training | Control/Unexposed
Number analyzed (Participants) | 28 | 27
score on a scale | 0.68 (2.29) | 1.13 (2.09)
Statistical Analysis 1: Comparison: Exposed to GRIN Training vs Control/Unexposed; Test type: Superiority; p = 0.39, Regression, Linear; Slope = -9.29, 95% CI 2-sided [-31.15 to 12.56], Standard Error of Mean 10.74

ADVERSE EVENTS:
Time Frame: Baseline to 2 weeks
Description: no adverse events measured
Arm/Group | Exposed to GRIN Training | Control/Unexposed
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/45
Other Adverse Events (participants affected / at risk) | 0/62 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT05511935/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT05511935/SAP_001.pdf